CLINICAL TRIAL: NCT06003634
Title: Older Adults Using Social Support to Improve Self-Care: Adaptation, Implementation, and Feasibility of Peer Support for Older Adults With T2DM in Appalachia.
Brief Title: OASIS: Peer Support for T2DM in Appalachia (Peer Coaches)
Acronym: OASIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brittany L Smalls (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Brittany L Smalls, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 83904; R01DK135885-01 (NIH)
Record Dates: First submitted 2023-07-31; First posted 2023-08-22 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Appalachian Region; Peer Influence; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Peer participants will be linked to a peer coach in one of four ways: (1) self-select coach with contact once a week (2) self-selected coach with contact every 2 weeks (3) matched with peer coach with contact once a week (4) matched with peer coach with contact every 2 weeks. Profile sheets that detail age, region of residence, hobbies etc. of each peer coach will be provided to peer participants who will then rank their top three choices. Matching will be completed by study personnel, and will be based mostly in region of residence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Peer Participants (A) (Experimental): Peer participants in group A will self select a peer coach using peer coach profile sheets, and will be contacted weekly during intervention period.
  Interventions: Behavioral: Peer Coaching - Peer Participants A
- Peer Participants (B) (Experimental): Peer participants in group B will self select a peer coach using peer coach profile sheets, and will be contacted weekly during intervention period.
  Interventions: Behavioral: Peer Coaching - Peer Participants B
- Peer Participants (C) (Experimental): Peer participants in group C will self select a peer coach using peer coach profile sheets, and will be contacted weekly during intervention period.
  Interventions: Behavioral: Peer Coaching - Peer Participants C
- Peer Participants (D) (Experimental): Peer participants in group D will self select a peer coach using peer coach profile sheets, and will be contacted weekly during intervention period.
  Interventions: Behavioral: Peer Coaching - Peer Participants D

INTERVENTIONS:
Behavioral: Peer Coaching - Peer Participants A — Peer participants in group A will self select a peer coach and will be contacted weekly by peer coaches.
  Arms: Peer Participants (A)
Behavioral: Peer Coaching - Peer Participants B — Peer participants in group B will self select a peer coach and will be contacted bi-weekly by peer coaches.
  Arms: Peer Participants (B)
Behavioral: Peer Coaching - Peer Participants C — Peer participants in group C will be matched with a peer coach and will be contacted weekly by peer coaches.
  Arms: Peer Participants (C)
Behavioral: Peer Coaching - Peer Participants D — Peer participants in group D will be matched with a peer coach and will be contacted bi-weekly by peer coaches.
  Arms: Peer Participants (D)

SUMMARY:
The goal of this clinical trial is to compare the effects of peer coaching models in older adults with unmanaged type two diabetes. The main questions it aims to answer are:

* Are peer coaching models effective at promoting Type 2 Diabetes Mellitus self-management?
* If effective, which facets of the peer model are most effective? Peer coaches will
* Undergo peer coach training.
* Reach out to peer participants on a weekly/biweekly time frame to discuss self-management and goal setting.
* Retain records of contact, topics discussed, and general notes on interactions. Researchers will compare differences in the frequency of contact, as well as how peer coaches were matched to peer participants to see if efficacy of the intervention is altered between groups.

DETAILED DESCRIPTION:
The Older Adults using Social Support to Improve Self-Care (OASIS) intervention is an asset-based approach, utilizing the unique social structure existing in Kentucky's rural Appalachian communities to address self-care behaviors as they relate to Type 2 Diabetes Mellitus (T2DM) management. The intervention will be composed of two groups: peer coaches who have managed T2DM (HbA1c < 7.5%), and peer participants who have unmanaged T2DM (HbA1c> 7.5%). Peer coaches will undergo training prior to intervention initiation to develop coaching skills. Peer participants will be linked to a peer coach in one of four ways: (1) self-select coach with contact once a week (2) self-selected coach with contact every 2 weeks (3) matched with peer coach with contact once a week (4) matched with peer coach with contact every 2 weeks. In addition to evaluating the effectiveness of a peer coaching model, the four groups will be evaluated allowing for a more detailed understanding of factors that influence self-care behaviors. Stakeholders will also be engaged at three time points: prior to the intervention, study mid-point, and at study conclusion. At study conclusion, a small cohort of both peer participants and peer coaches will be invited to contribute to stakeholder group interviews. Information exchange with stakeholders will aid in developing a robust understanding of influential factors and how to effectively promulgate the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 55 years
* Resident in Rural Kentucky
* Positive diagnosis of Type 2 Diabetes Mellitus
* HbA1c less than 7.5 for peer coaches
* Passing score on cognitive assessment administered by study personnel
* English Speaking

Exclusion Criteria:

* Age less than 55 years
* Not a resident of a Rural Kentucky county
* Cognitive Impairment
* Non-English Speaking

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Change in A1c | Collected at Baseline, 3 month, and 6 month follow up.
  Obtained using Point of Care assessment

SECONDARY OUTCOMES:
Diabetes Empowerment | Collected at Baseline, 3 month, and 6 month follow up.
  "Attitudes Towards Diabetes- DES". 5 point scale ranging from 1 "Strongly Agree" to 5 "Strongly Disagree", where lower scores indicate greater feelings of empowerment.
Quality of Life Index | Collected at Baseline, 3 month, and 6 month follow up.
  "EuroQofL-5D" measures acts of daily living (ADL) on a five point scale ranging from 0 "no" problems to 5 "extreme" problems, where higher scores indicate lower ability to engage in ADL.
Social Support | Collected at Baseline, 3 month, and 6 month follow up.
  "MOS Social Support Survey" a five point scale ranging from 1 "none of the time" to 5 "all of the time" where higher scores indicate better social support.
Depression Scale | Collected at Baseline, 3 month, and 6 month follow up.
  "Geriatric Depression Scale: Short Form" is a binary survey where participants can select "yes" or "no". Each "yes" is a singular point, if a score >5 points it is suggestive about depression and warrant a follow-up comprehensive assessment. A score of greater than or equal to 10 is almost always indicative of depression.
Problem Areas in Diabetes | Collected at Baseline, 3 month, and 6 month follow up.
  "Problem Areas In Diabetes (PAID) Scale" a five point scale ranging from 0 "not a problem" to 4 "serious problem", where a higher score indicates more problems in diabetes management.
Diabetes Self-Management | Collected at Baseline, 3 month, and 6 month follow up.
  Diabetes Self-Management Questionnaire (DSMQ) is a four point scale ranging from 0 "does not apply to me" to 3 "applies to me very much". Higher scores indicate better diabetes management.
Acts of Daily Living | Collected at Baseline, 3 month, and 6 month follow up.
  "Lawton-Brody Instrumental Activities of Daily Living Scale (L.A.D.L) is a binary where "0" is low functioning and "1" is high functioning. Higher scores indicate higher functioning.
Social Network Scale | Collected at Baseline, 3 month, and 6 month follow up.
  "Lubbens Social Network Scale - 6 (LSNS-6) is a five point scale ranging from "0" none to "5" nine or more. Higher scores indicate greater amount of social support.

CONTACTS AND LOCATIONS:
Overall Officials: Brittany L Smalls, PhD, Principal Investigator — University of Kentucky
Locations (2):
- United States (2):
  - Barren River Area Development District, Bowling Green, Kentucky
  - UK HealthCare, Hazard, Kentucky

REFERENCES:
- [Derived] Smalls BL, Kruse-Diehr A, Ortz CL, Douthitt K, McLouth C, Shelton R, Taylor Z, Williams E. Older adults using social support to improve self-care (OASIS): Adaptation, implementation and feasibility of peer support for older adults with T2D in appalachia: A feasibility study protocol. PLoS One. 2024 Mar 18;19(3):e0300196. doi: 10.1371/journal.pone.0300196. eCollection 2024. PMID 38498512